CLINICAL TRIAL: NCT01411670
Title: Administration of Human Protein C Concentrates in Patients With Sepsis and Septic Shock: Effects on Microcirculation and Organ Function.
Brief Title: Administration of Human Protein C Concentrates in Patients With Sepsis and Septic Shock.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Andrea Morelli, associate professor, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2112
Record Dates: First submitted 2011-08-05; First posted 2011-08-08 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-12

CONDITIONS: Sepsis; Septic Shock
Keywords: Human Protein C; Activated protein C; Microcirculation; Septic Shock; Sepsis
MeSH Terms: conditions — Sepsis; Shock, Septic | interventions — Protein C

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Human protein C concentrate (Experimental)
  Interventions: Drug: Human protein C concentrate
- activated protein C (Active Comparator): Continuous infusion of Activated Protein C
  Interventions: Drug: Activated protein C
- Placebo (Placebo Comparator): Standard treatment
  Interventions: Drug: Placebo comparator

INTERVENTIONS:
Drug: Human protein C concentrate — Continuous infusion of human protein C concentrate at the dose of 3 UI/Kg/Hr to reach a protein C plasma activity of 70-120%
  Arms: Human protein C concentrate
Drug: Activated protein C — Continuous infusion of activated protein C at the dose of 24 micrograms/Kg/Hr for 96 hours
  Arms: activated protein C
Drug: Placebo comparator — Standard treatment
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the effects on systemic hemodynamics, microcirculation and organ function of human Protein C concentrate in patients with sepsis and septic shock.

DETAILED DESCRIPTION:
Sixty septic patients with plasma protein C activity < 60 % will be enrolled in the study. Patients will be randomly allocated to be treated with either a) a continuous infusion of human Protein C concentrate at 3 UI/Kg/hr for 72 hours to reach plasma protein C activity between 70 and 120 % b)to a continuous infusion of activated protein C at 24 micrograms/Kg/hr for 96 hours, c) a standard teatment(control; each n = 20). In all groups, norepinephrine will be titrated to achieve a mean arterial pressure (MAP) between 65 and 75 mmHg. Data from right heart catheterization, from microcirculation (SDF imaging) and from organ function as well as norepinephrine requirements will be obtained at baseline and after 24, 48, 72 hours.

ELIGIBILITY:
Inclusion Criteria:

* Severe sepsis or septic shock with plasma activity of protein C < 60 %

Exclusion Criteria:

* Pregnancy
* Risk of Bleeding
* Hemorragia
* age < 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-01; Primary Completion 2015-02 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
plasma protein C activity | over a period of 72 hours

SECONDARY OUTCOMES:
sublingual microcirculatory blood flow | over a period of 72 hours
  Systemic hemodynamics,sublingual microcirculatory blood flow, organ function, citokynes.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Morelli, MD, Principal Investigator — University of Roma La Sapienza
Locations (1):
- Departement of Anesthesiology and Intensive Care of the University of Rome La Sapienza, Rome, Italy